CLINICAL TRIAL: NCT00002063
Title: Treatment of AIDS and AIDS Related Complex. Part-1- Treatment of Patients With ARC (AZT Vs. Placebo)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 016A; VA Study 298
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-01

CONDITIONS: HIV Infections
Keywords: Immune Tolerance; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
Primary: To determine the clinical effect of zidovudine (AZT) compared to placebo in terms of time to progression to AIDS (i.e., occurrence of major opportunistic infections, dementia, and malignancies) or death. Initial drug assignment will be changed to open-label AZT for patients who experience a sustained decline in CD4 lymphocyte concentration to less than 200 cells/mm3, but analysis will be based on initial treatment assignment. To determine the immunologic effect of AZT compared to placebo in terms of time to drop in CD4 lymphocyte concentration of at least 25 percent from baseline assessment. To determine the antiviral effect of AZT compared to placebo in eradicating or suppressing HIV. Secondary: To determine the effect of AZT compared to placebo on the immune status of HIV-infected patients by comparing lymphocyte profiles and indices. To determine the long-term toxicities of AZT compared to placebo in terms of abnormalities in BL, hepatic function, renal function, skin, gastrointestinal system, and central nervous system. To describe the natural history of AIDS related complex (ARC) in placebo patients in terms of initial CD4 lymphocyte concentration and the Walter Reed staging system.

ELIGIBILITY:
Inclusion Criteria

Patient must have AIDS related complex (ARC) as defined by Walter Reed stages, be ambulatory, and be able to give informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with unstable disease characterized by the following are excluded:

* Hospitalization within the past 14 days.
* Major opportunistic infection, current or past.
* An active infection of onset during the past 30 days, as evidenced by symptoms, signs, or laboratory abnormalities such as:
* Temperature = or > 100.5 degrees F.
* Night sweats.
* Weight loss = or > 10 percent of body weight.
* Diarrhea (3 or more bowel movements/day).
* Persistent cough, shortness of breath, or dyspnea on exercise.
* Abnormal chest x-ray suggesting pneumonia or increased arterial-alveolar (A-a) gradient.
* Altered mental status, seizures, or focal neurologic signs.
* Abnormal computerized tomography (CT) scan or magnetic resonance imaging (MRI) suggestive of toxoplasmosis, peripheral mononuclear leukocytes, lymphoma, or other focal abnormality of the central nervous system (CNS).
* Abnormal cerebrospinal fluid (CSF) suggestive of cryptococcal, mycobacterial, or other meningitis. (The decision to perform invasive tests, such as lumbar puncture, specialized microbiological tests such as bone marrow culture for Mycobacteria or Histoplasma capsulatum, or specialized radiological tests such as CT scan or MRI should be based on clinical assessment of the patient.)
* Kaposi's sarcoma.
* Lymphoma; malignancy requiring chemotherapy.
* Dementia.
* Requiring hemodialysis or renal insufficiency or failure.
* Leukopenia.
* Thrombocytopenia.

Patients with the following are excluded:

* Unstable disease.
* Kaposi's sarcoma.
* Lymphoma; malignancy requiring chemotherapy.
* Dementia.
* Major opportunistic infection, current or past.
* Anemia (hemoglobin less than 9.5 g/dl).

Prior Medication:

Excluded within 1 month of study entry:

* Ribavirin or zidovudine (AZT) or other antivirals.
* Immunomodulating agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Wadsworth Veterans Administration Med Ctr, Los Angeles, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Walter Reed Army Med Ctr, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - Dr Gordon Dickinson, Miami, Florida
  - Dr Gigi Diamond / New York Veterans Administration, New York, New York
  - Veterans Affairs Med Ctr / Admin Only / Not For Patient Care, Durham, North Carolina
  - Houston Veterans Administration Med Ctr, Houston, Texas